CLINICAL TRIAL: NCT00549913
Title: A Dose-escalation Study to Assess the Feasibility and Safety of 3 Different Doses of NeoFuse When Combined With MasterGraft Granules in Subjects Requiring Posterolateral Lumbar Fusion With Instrumentation.
Brief Title: Study of 3 Doses of NeoFuse Combined With MasterGraft Granules in Subjects Requiring Posterolateral Lumbar Fusion (PLF)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSF0106
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Spinal Stenosis
Keywords: adjacent vertebral levels between L1 and S1
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Spinal Stenosis | interventions — Spinal Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): 10 subjects to receive lowest dose of NeoFuse (MPCs)
  Interventions: Biological: NeoFuse
- 2 (Active Comparator): 4 subjects standard posterolateral spinal fusion with instrumentation
  Interventions: Procedure: posterolateral spinal fusion with instrumentation
- 3 (Experimental): 10 subjects to receive middle dose of NeoFuse
  Interventions: Biological: NeoFuse
- 4 (Active Comparator): 3 subjects standard posterolateral spinal fusion with instrumentation
  Interventions: Procedure: posterolateral spinal fusion with instrumentation
- 5 (Experimental): 10 subjects to receive highest dose of NeoFuse
  Interventions: Biological: NeoFuse
- 6 (Active Comparator): 3 subjects with standard posterolateral spinal fusion with instrumentation
  Interventions: Procedure: posterolateral spinal fusion with instrumentation

INTERVENTIONS:
Biological: NeoFuse — immunoselected, culture-expanded, nucleated, allogeneic MPCs (NeoFuse) combined with MasterGraft Resorbable Ceramic Granules in subjects requiring posterior lumbar interbody fusion with NuVasive's radiolucent PEEK OPTIMA cage
  Other Names: Spinal Fusion; Stem Cells
  Arms: 1; 3; 5
Procedure: posterolateral spinal fusion with instrumentation — autograft in subjects requiring posterior lumbar interbody fusion with NuVasive's radiolucent PEEK OPTIMA cage
  Other Names: Spinal Fusion; Controls
  Arms: 2; 4; 6

SUMMARY:
This is a first-in-human, dose escalation clinical study to evaluate the feasibility, safety, and tolerability of 3 different doses of immunoselected, culture-expanded, nucleated, allogeneic MPCs (NeoFuse) when combined with MasterGraft Resorbable Ceramic Granules (Medtronic Sofamor Danek USA, Inc.) compared to autograft in patients requiring posterior lumbar interbody fusion with NuVasive's radiolucent PEEK OPTIMA cage (to be used with autologous bone graft material) and 1 or 2 level posterolateral lumbar fusion surgery with instrumentation. The instrumentation used for this study will be the Monarch® 5.50 mm Spine System (DePuy).

DETAILED DESCRIPTION:
This is a prospective, single center, randomized, open-label controlled Phase 1b/2a study designed to evaluate the safety and preliminary efficacy of MPCs combined with MasterGraft Granules when compared to use of autologous bone graft in the posterolateral fusion site in subjects requiring interbody fusion in combination with instrumented 1 or 2 level PLF procedure. All subjects in this study will undergo a 1 or 2-level (2 or 3 vertebrae) interbody fusion without the use of the investigational product.

In addition to the interbody fusion procedure, subjects will undergo an instrumented posterolateral fusion. NeoFuse plus MasterGraft Granules at one of three doses or autograft will be implanted in the posterolateral lumbar fusion site(s) only.

After the screening and surgical visits, each subject will be evaluated clinically and radiographically within 3 days and 30 days after surgery, and at 3, 6, and 12 months after surgery.

Subjects will be evaluated at 24 and 36 months after surgery for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. Have a documented symptomatic diagnosis of DDD at L1-S1 with or without stenosis and with or without up to and including Grade II degenerative spondylolisthesis.
3. May also have coexistent spinal or foraminal stenosis as confirmed by MRI or CT evaluation.
4. Must have clinical symptoms of neurogenic claudication.
5. Must have failed 6 months of nonoperative management.
6. Must be a candidate for lumbar interbody fusion in combination with posterolateral lumbar fusion with the use of autograft from the iliac crest requiring a 1 or 2-level fusion of adjacent vertebral levels between L1 and S1.
7. Must have a stable screening electrocardiogram (ECG), as determined by the investigator that would not preclude surgery.

Exclusion Criteria:

1. Is pregnant or breastfeeding.
2. Has Grade III or greater spondylolisthesis.
3. Has or is undergoing revision of a prior fusion at the involved levels.
4. Has a history of hypersensitivity or anaphylactic reaction to murine or bovine products, dimethyl sulfoxide (DMSO), or titanium.
5. Has MRI or CT that shows greater than 50% anterior translocation of cranial vertebral body or greater than 20 degree angular motion of the listhesis segment.
6. Has a history of active malignancy in the last 5 years, other than basal cell carcinoma.
7. Has osteoporosis as defined by a dual energy x-ray absorptiometry (DXA T) score of ≤ -3.5 or a history of fragility fractures or other significant bone disease contraindicating the use of spinal instrumentation.

   Note: subjects will be screened using the Simple Calculated Osteoporosis Risk Evaluation (SCORE) osteoporosis questionnaire.
8. Has a history of Paget's disease of the spine, osteomalacia, or any other metabolic bone disease.
9. Has a history of prior radiotherapy to the involved area.
10. Has received systemic corticosteroids at a dose equivalent to prednisone > 10 mg/day within 14 days prior to study procedure.
11. Has received systemic nonsteroidal anti-inflammatory drugs (NSAIDS) within 48 hours prior to study procedure, and unwilling to refrain from NSAIDS for the first 6 months following the procedure.
12. Has a positive screen for human immunodeficiency virus (HIV) antibodies.
13. Has had treatment with any investigational therapy administered within 6 months before implantation surgery. .
14. Is the prior recipient of allogeneic stem cell/progenitor cell therapy.
15. Has a body mass index (BMI) > 3.5
16. Has 20% or greater anti-human leukocyte antigen (HLA) antibody titer and/or has antibody specificities to donor HLA antigens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-10; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety of NeoFuse (allogeneic mesenchymal precursor cells [MPCs]) when combined with MasterGraft Resorbable Ceramic Granules as a carrier for posterolateral lumbar fusion with instrumentation. | 30 days

SECONDARY OUTCOMES:
To evaluate the overall fusion success of the use of NeoFuse plus carrier compared to autograft in the same patient | 3 years
To assess CT scan as a pilot measure of fusion for use in the pivotal study | 3 years
To provide preliminary data to support dose selection | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Donna Skerrett, MD, Study Director — Mesoblast, Ltd.
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- See also: The Sponsor's web site — http://www.mesoblast.com